CLINICAL TRIAL: NCT05698108
Title: Effects Of Instrument Assisted Soft Tissue Mobilization Using Ergon Technique on Pain, Grip Strength and Functional Activity in Patients With Lateral Epicondylitis: A Randomized Controlled Trial
Brief Title: Effects Of Instrument Assisted Soft Tissue Mobilization on Pain, Grip Strength and Functional Activity in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULahore Shazal Nazir
Record Dates: First submitted 2022-11-26; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: IASTM; Lateral Epicondylitis; tennis elbow; pain; grip strength; functional activity
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The study was single-blinded as the assessor was blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physcial Therapy Group (Active Comparator): All participants received treatment 2 times a week for 4 weeks. Pre-treatment included a Moist hot pack for 10 minutes and traditional physical therapy included Cyriax Deep Friction Massage (DFM), Ultrasound therapy as well as strengthening and stretching exercises
  Interventions: Other: Conventional Physical Therapy
- IASTM Group (Experimental): Participants received Instrument Assisted Soft Tissue Mobilization Treatment 2 times a week for 4 weeks using Ergon IASTM tools.
  Interventions: Device: Instrument Assisted Soft Tissue Mobilization (IASTM)

INTERVENTIONS:
Device: Instrument Assisted Soft Tissue Mobilization (IASTM) — Tools designed for soft tissue mobilization
  Other Names: Ergon Tools
  Arms: IASTM Group
Other: Conventional Physical Therapy — Moist Hot pack, Ultrasound, Deep Friction Massage, Stretching and Strengthening Exercises.
  Other Names: Traditional Physical Therapy
  Arms: Conventional Physcial Therapy Group

SUMMARY:
This study aimed to find the effects of Instrument Assisted Soft Tissue Mobilization (IASTM) using Ergon Tools on pain, grip strength and functional activity among patients diagnosed with Lateral epicondylitis.

The study concluded that IASTM is effective in improving pain, grip strength and functional activity in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
Background: Lateral Epicondylitis is a type of "repetitive strain injury" that causes pain on the lateral portion of the elbow, especially while gripping and applying resistance to the forearm's extensor muscles, both men and women are equally affected by it. Traditional Physical Therapy has failed to improve the disorders caused by LE, Instrument Assisted Soft Tissue Mobilization is a new approach for its treatment a lot of tools are being used and Ergon Tools are among one of them, very less data is available for its efficacy in lateral epicondylitis patients.

Objective: To compare the effects of Instrument Assisted Soft Tissue Mobilization using Ergon Technique on pain, grip strength and functional activity in patients with lateral epicondylitis.

Methodology: 72 individuals with lateral epicondylitis pre-diagnosed by an orthopedic surgeon, are assessed from Sikander Medical Complex, Gujranwala. After fulfilling the inclusion criteria, the participants are randomly divided into two groups, 36 participants receiving IASTM using Ergon Tools and 36 participants received conventional physical therapy. Both groups receive treatment 2 times a week for 4 weeks. Outcome measures are pain (VAS), grip strength (handheld dynamometer), and functional mobility (PRTEE) collected at the baseline, 1st week, and 4th week.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female Patients
* Patients between the age group 20-50 years
* Sub-acute Patients having symptoms for > 6 weeks and < 3 months.
* Patients who had pain rating from 5 to 9 in VAS will be included
* Patients with Positive Cozens test, Mill's test

Exclusion Criteria:

* Patients with any surgical or trauma history of the elbow
* Rheumatoid Arthritis and Malignancies
* Cervical Radiculopathy patients who have referred pain in the elbow
* Loss of Passive ROM in extension
* Active infections such as, Bursitis, Calcification of the soft tissues, Fragile skin, Hyper Mobility & Joint Effusion
* Hemophilic Patients
* Osteoporosis
* Patients with history of getting treatment with Steroid Injections will be excluded.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Pain (mild to severe) | 4 weeks
  Visual Analogue Scale The score is calculated by measuring the distance (mm) between the "no pain" anchor and the patient's mark on a 10-cm line with a ruler, yielding a range of 0-100. A higher score implies that the pain is more intense and a lower score suggests the intensity of pain to be milder. VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain
Grip Strength | 4 weeks
  Digital Hand Held Dynamometer The best result from several trials for each hand is recorded, with at least 15 seconds recovery between each effort. The values listed below (in kg and lbs) give a guide to expected scores for adults. These values are the average of the best scores of each hand. See more Hand Grip Strength Norms. Other protocols will just use the score from the dominant hand, or compare the left and right hand results. See also examples of some actual athlete results.
Functional Activity | 4 weeks
  Patient Rated Tennis Elbow Evaluation It consists of pain subscale and functional subscale, total score is calculated by adding Pain Subscale and Function Subscale then calculated as, Best Score= 0 Worst Score = 100 (pain and disability contribute equally to score)

CONTACTS AND LOCATIONS:
Overall Officials: Shazal Nazir, DPT, Principal Investigator — University of Lahore
Locations (1):
- Sikander Medical Complex, Gujranwala, Pujab, Pakistan